CLINICAL TRIAL: NCT01515956
Title: A Phase 2, Open-label, Multinational Clinical Study to Evaluate the Safety and Efficacy of BMN 110 in Pediatric Patients Less Than 5 Years of Age With Mucopolysaccharidosis IVA (Morquio A Syndrome)
Brief Title: Study of BMN 110 in Pediatric Patients < 5 Years of Age With Mucopolysaccharidosis IVA (Morquio A Syndrome)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BioMarin Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MOR-007
Record Dates: First submitted 2011-12-22; First posted 2012-01-24 (Estimated); Results first posted 2017-07-06 (Actual); Last update posted 2017-08-10 (Actual); Status verified 2017-07

CONDITIONS: Mucopolysaccharidosis IVA; Morquio A Syndrome; MPS IVA
Keywords: Mucopolysaccharidosis IVA type A; MPS IVA Type A; Mucopolysaccharidosis IVA; MPS IVA; Morquio A Syndrome; Lysosomal Storage Disorder; LSD; N-acetylgalactosamine-6-sulfatase; N-acetylgalactosamine-6-sulfate; sulfatase; galactose-6-sulfatase; GALNS; enzyme replacement therapy; ERT
MeSH Terms: conditions — Mucopolysaccharidosis IV; Lysosomal Storage Diseases | interventions — GALNS protein, human; Chondroitinases and Chondroitin Lyases; Galns protein, mouse; Sulfatases; Enzyme Replacement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- BMN 110 Weekly (Experimental)
  Interventions: Drug: BMN 110

INTERVENTIONS:
Drug: BMN 110 — Patients will receive intravenous (IV) infusions of study drug at a dose of 2.0 mg/kg/wk over a period of approximately 4 hours every week for up to 208 weeks.
  Other Names: N-acetylgalactosamine-6-sulfatase; N-acetylgalactosamine-6-sulfate; sulfatase; galactose-6-sulfatase; GALNS; enzyme replacement therapy; ERT

SUMMARY:
This open-label Phase 2 study will evaluate the safety and efficacy of weekly 2.0 mg/kg/wk infusions of BMN 110 in pediatric patients, less than 5 years of age at the time of administration of the first dose of study drug, diagnosed with MPS IVA (Morquio A Syndrome) for up to 208 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Less than 5 years of age at the time of the first study drug infusion
* Documented clinical diagnosis of MPS IVA based on clinical signs and symptoms of MPS IVA and documented reduced fibroblast or leukocyte GALNS enzyme activity or genetic testing confirming diagnosis of MPS IVA
* Written informed consent provided by parent or legally authorized representative after the nature of the study has been explained and prior to any research-related procedures.

Exclusion Criteria:

* Previous hematopoietic stem cell transplant (HSCT).
* Previous treatment with BMN 110.
* Known hypersensitivity to any of the components of BMN 110.
* Major surgery within 3 months prior to stuy entry or planned major surgery during the 52-week treatment period.
* Use of any investigational product or investigational medical device within 30 days prior to Screening, or requirement for any investigational agent prior to completion of all scheduled study assessments.
* Concurrent disease or condition, including but not limited to symptomatic cervical spine instability, clinically significant spinal cord compression, or severe cardiac disease that would interfere with study participation or safety as determined by the Investigator.
* Any condition that, in the view of the Investigator, places the subject at high risk of poor treatment compliance or of not completing the study.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2011-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Lounsbury, Study Director — BioMarin Pharmaceutical
Locations (5):
- United States (2):
  - Oakland, California
  - Manhasset, New York
- Monza, Italy
- Taipei, Taiwan
- Central Manchester, United Kingdom

REFERENCES:
- [Derived] Jones SA, Bialer M, Parini R, Martin K, Wang H, Yang K, Shaywitz AJ, Harmatz P. Safety and clinical activity of elosulfase alfa in pediatric patients with Morquio A syndrome (mucopolysaccharidosis IVA) less than 5 y. Pediatr Res. 2015 Dec;78(6):717-22. doi: 10.1038/pr.2015.169. Epub 2015 Sep 2. PMID 26331768

RESULTS

PARTICIPANT FLOW:
Groups:
- BMN110 2.0 mg/kg/Week: Weekly intravenous infusions of BMN 110 at a dose of 2.0 mg/kg for 52 consecutive weeks. Each infusion will be administered over a period of approximately 4 hours.
Period: Overall Study
Arm/Group | BMN110 2.0 mg/kg/Week
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- BMN110 2.0 mg/kg/Week: 2.0 mg/kg/week
Arm/Group | BMN110 2.0 mg/kg/Week
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.1 (1.34)
Age, Customized [Number; unit: participants]
  0 to <3 years | 7
  >=3 to <5 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 4
  White | 10
  Other | 1
Region of Enrollment [Number; unit: participants]
  Italy | 2
  United Kingdom | 6
  United States | 7
Urinary Keratan Sulfate Measures [Mean (Standard Deviation); unit: ug/mg] | 35.9 (12.32)

OUTCOME MEASURES:

1. Primary Outcome: To Evaluate Safety and Tolerability of Infusions of BMN 110 at a Dose of 2.0 mg/kg/Week Over a 52-week Period in MPS IVA Subjects Less Than 5 Years of Age at Time of First Study Drug Infusion
Description: Number of Participants Experiencing Adverse Events
Time Frame: 52 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- BMN110 2.0 mg/kg/Week: BMN110 2.0 mg/kg/week
Arm/Group | BMN110 2.0 mg/kg/Week
Number analyzed (Participants) | 15
Participants | 15

2. Secondary Outcome: Percent Change From Baseline to Week 52 in Urinary Keratan Sulfate Measures
Description: Percent Change from Baseline to Week 52 for Urinary Keratan Sulfate measures.
Time Frame: Baseline to Week 52
Population: Efficacy Analysis Set - All enrolled patients with at least 1 post treatment efficacy measurement will be included in efficacy analyses.
Measure: Mean (Standard Deviation); unit: percentage change
Arm/Group | BMN110 2.0 mg/kg/Week
Number analyzed (Participants) | 11
percentage change | -44.3 (21.15)

3. Secondary Outcome: Change From Baseline in Normalized Growth Rate Z-Scores
Description: Changes in growth over time will be assessed using anthropometric measurements and radiographs of lower extremities. Z-scores are the normalized scores derived from the reference population mean and standard deviation (A positive change from baseline indicates that the population has moved closer to the reference population and represents a positive outcome).
Time Frame: Baseline to Week 52
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: z-score
Arm/Group | BMN110 2.0 mg/kg/Week
Number analyzed (Participants) | 15
z-score
  Baseline: number analyzed (Participants) | 8
  Baseline | -0.6 (0.64)
  Change from Baseline to Week 52: number analyzed (Participants) | 8
  Change from Baseline to Week 52 | 0.2 (1.04)

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | BMN110 2.0 mg/kg/Week
Serious Adverse Events (participants affected / at risk) | 8/15
Other Adverse Events (participants affected / at risk) | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN110 2.0 mg/kg/Week (N=15)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Medical device complication (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Joint instability (Musculoskeletal and connective tissue disorders) | 1 (1)
Knee deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebrospinal fluid leakage (Nervous system disorders) | 1 (1)
Cervical cord compression (Nervous system disorders) | 4 (4)
Spinal cord oedema (Nervous system disorders) | 1 (1)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Poor venous access (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BMN110 2.0 mg/kg/Week (N=15)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 4 (9)
Developmental hip dysplasia (Congenital, familial and genetic disorders) | 1 (1)
Aural polyp (Ear and labyrinth disorders) | 1 (1)
Cerumen impaction (Ear and labyrinth disorders) | 1 (1)
Conductive deafness (Ear and labyrinth disorders) | 1 (2)
Deafness (Ear and labyrinth disorders) | 2 (2)
Deafness bilateral (Ear and labyrinth disorders) | 1 (1)
Ear haemorrhage (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 3 (17)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Middle ear effusion (Ear and labyrinth disorders) | 1 (1)
Motion sickness (Ear and labyrinth disorders) | 1 (1)
Otorrhoea (Ear and labyrinth disorders) | 2 (2)
Amblyopia (Eye disorders) | 1 (1)
Astigmatism (Eye disorders) | 1 (1)
Conjunctivitis (Eye disorders) | 4 (5)
Conjunctivitis allergic (Eye disorders) | 1 (3)
Corneal opacity (Eye disorders) | 3 (3)
Eye discharge (Eye disorders) | 1 (3)
Eye pain (Eye disorders) | 1 (1)
Eye swelling (Eye disorders) | 2 (2)
Keratitis (Eye disorders) | 1 (1)
Trichiasis (Eye disorders) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 2 (4)
Abdominal pain (Gastrointestinal disorders) | 8 (14)
Abdominal pain upper (Gastrointestinal disorders) | 5 (14)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Dental caries (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 11 (24)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (2)
Gastritis (Gastrointestinal disorders) | 2 (3)
Gingival pain (Gastrointestinal disorders) | 1 (2)
Mouth ulceration (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 4 (5)
Oral discomfort (Gastrointestinal disorders) | 1 (1)
Oral disorder (Gastrointestinal disorders) | 1 (2)
Retching (Gastrointestinal disorders) | 1 (2)
Toothache (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 13 (59)
Catheter site extravasation (General disorders) | 4 (6)
Catheter site pain (General disorders) | 1 (1)
Catheter site related reaction (General disorders) | 2 (2)
Chest pain (General disorders) | 1 (1)
Chills (General disorders) | 1 (1)
Crepitations (General disorders) | 1 (1)
Device difficult to use (General disorders) | 1 (1)
Fatigue (General disorders) | 4 (6)
Gait disturbance (General disorders) | 1 (1)
Implant site haemorrhage (General disorders) | 1 (1)
Infusion site extravasation (General disorders) | 2 (3)
Injection site hypersensitivity (General disorders) | 1 (1)
Local swelling (General disorders) | 1 (1)
Malaise (General disorders) | 3 (4)
Mass (General disorders) | 1 (1)
Medical device complication (General disorders) | 1 (1)
Medical device pain (General disorders) | 1 (1)
Medical device site reaction (General disorders) | 1 (2)
Pain (General disorders) | 3 (3)
Pyrexia (General disorders) | 15 (143)
Hepatic function abnormal (Hepatobiliary disorders) | 1 (2)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1)
Acute sinusitis (Infections and infestations) | 1 (1)
Acute tonsillitis (Infections and infestations) | 1 (1)
Anal fungal infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 3 (7)
Conjunctivitis infective (Infections and infestations) | 1 (1)
Diarrhoea infectious (Infections and infestations) | 1 (1)
Ear infection (Infections and infestations) | 3 (4)
Exanthema subitum (Infections and infestations) | 1 (2)
Fungal skin infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 2 (3)
Gastroenteritis viral (Infections and infestations) | 1 (2)
Gingival infection (Infections and infestations) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 1 (1)
Herpes simplex (Infections and infestations) | 1 (2)
Hordeolum (Infections and infestations) | 1 (1)
Implant site infection (Infections and infestations) | 3 (3)
Influenza (Infections and infestations) | 3 (3)
Lower respiratory tract infection (Infections and infestations) | 2 (4)
Molluscum contagiosum (Infections and infestations) | 1 (2)
Nasopharyngitis (Infections and infestations) | 9 (25)
Oral candidiasis (Infections and infestations) | 1 (1)
Otitis externa (Infections and infestations) | 2 (2)
Otitis media (Infections and infestations) | 5 (6)
Otitis media acute (Infections and infestations) | 3 (6)
Otitis media chronic (Infections and infestations) | 1 (1)
Penile infection (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 2 (3)
Postoperative wound infection (Infections and infestations) | 1 (1)
Rash pustular (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 9 (22)
Skin infection (Infections and infestations) | 2 (2)
Tonsillitis (Infections and infestations) | 1 (1)
Tooth infection (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 8 (52)
Urinary tract infection (Infections and infestations) | 1 (2)
Viral infection (Infections and infestations) | 2 (2)
Viral rash (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 5 (8)
Contusion (Injury, poisoning and procedural complications) | 5 (5)
Eye contusion (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (3)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (3)
Injury corneal (Injury, poisoning and procedural complications) | 1 (1)
Laceration (Injury, poisoning and procedural complications) | 1 (2)
Limb crushing injury (Injury, poisoning and procedural complications) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1)
Postoperative fever (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1)
Scar (Injury, poisoning and procedural complications) | 1 (1)
Spinal cord injury (Injury, poisoning and procedural complications) | 1 (1)
Thermal burn (Injury, poisoning and procedural complications) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Blood bicarbonate decreased (Investigations) | 2 (2)
Body temperature increased (Investigations) | 3 (5)
Breath sounds abnormal (Investigations) | 1 (1)
Heart rate increased (Investigations) | 3 (11)
Oxygen saturation decreased (Investigations) | 1 (1)
Respiratory rate increased (Investigations) | 2 (10)
Venous pressure decreased (Investigations) | 2 (2)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 (15)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Joint swelling (Musculoskeletal and connective tissue disorders) | 1 (1)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (15)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebral haematoma (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 5 (13)
Hypoaesthesia (Nervous system disorders) | 1 (2)
Agitation (Psychiatric disorders) | 2 (3)
Dysuria (Renal and urinary disorders) | 2 (2)
Haematuria (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Vesicoureteric reflux (Renal and urinary disorders) | 1 (1)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1)
Oedema genital (Reproductive system and breast disorders) | 1 (1)
Adenoidal hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Allergic respiratory disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (39)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Laryngospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (15)
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4 (23)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 8 (20)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 3 (5)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 2 (3)
Cold sweat (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (3)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 2 (2)
Eczema (Skin and subcutaneous tissue disorders) | 4 (5)
Erythema (Skin and subcutaneous tissue disorders) | 3 (3)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (7)
Rash (Skin and subcutaneous tissue disorders) | 6 (9)
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Skin reaction (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 4 (36)
Catheter placement (Surgical and medical procedures) | 1 (1)
Central venous catheter removal (Surgical and medical procedures) | 1 (1)
Central venous catheterisation (Surgical and medical procedures) | 2 (2)
Dental care (Surgical and medical procedures) | 1 (1)
Ear tube insertion (Surgical and medical procedures) | 1 (1)
Ear tube removal (Surgical and medical procedures) | 1 (1)
Infusion (Surgical and medical procedures) | 1 (1)
Joint fluid drainage (Surgical and medical procedures) | 1 (1)
Orchidopexy (Surgical and medical procedures) | 1 (1)
Flushing (Vascular disorders) | 3 (3)
Hot flush (Vascular disorders) | 1 (1)
Hyperaemia (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 2 (2)
Pallor (Vascular disorders) | 1 (1)
Poor venous access (Vascular disorders) | 4 (6)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes